CLINICAL TRIAL: NCT00016341
Title: Randomized Phase III Crossover Trial of Chemotherapy (Doxorubicin/Cisplatin/Paclitaxel and G-CSF) Versus Hormonal Therapy (Tamoxifen/Megestrol Acetate) in Patients With Stage III & IV or Recurrent Endometrial Cancer
Brief Title: Combination Chemotherapy Compared With Hormone Therapy in Treating Patients With Recurrent, Stage III, or Stage IV Endometrial Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068624; GOG-0189
Record Dates: First submitted 2001-05-06; First posted 2003-09-09 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2007-06

CONDITIONS: Endometrial Cancer
Keywords: stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Filgrastim; Cisplatin; Doxorubicin; Megestrol Acetate; Paclitaxel; Tamoxifen

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: megestrol acetate
Drug: paclitaxel
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Estrogen can stimulate the growth of tumor cells. Hormone therapy using tamoxifen and megestrol may fight endometrial cancer by blocking the absorption of estrogen. It is not yet known whether chemotherapy is more effective than hormone therapy in treating endometrial cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with that of hormone therapy in treating patients who have recurrent, stage III, or stage IV endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free survival and response of patients with stage III or IV or recurrent endometrial cancer treated with doxorubicin, cisplatin, paclitaxel, and filgrastim (G-CSF) vs tamoxifen and megestrol.
* Compare the survival of patients treated with these regimens.
* Determine if progesterone receptor status provides information on whether patients are more likely to benefit from chemotherapy.
* Compare the toxicity profiles of these treatment regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, cross-over, multicenter study. Patients are stratified according to progesterone receptor status (negative vs positive). Patients are randomized to 1 of 2 treatment arms.

* Arm I:Patients receive chemotherapy comprising doxorubicin IV over 15-30 minutes followed by cisplatin IV over 1 hour on day 1; paclitaxel IV over 3 hours on day 2; and filgrastim (G-CSF) subcutaneously beginning on day 3 and continuing for 10 days. Chemotherapy repeats every 21 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.
* At time of disease progression, patients cross-over to hormonal therapy as in arm II.
* Arm II: Patients receive hormonal therapy comprising oral megestrol twice daily on weeks 1-3 followed by oral tamoxifen twice daily on weeks 4-6. Hormonal therapy repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

At time of disease progression, if patients have not previously been enrolled on arm I, patients cross-over to receive chemotherapy as in arm I.

Quality of life is assessed at baseline, 6 weeks, time of progression, and then after 6 weeks on cross-over therapy.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 630 patients will be accrued for this study within 42 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary stage III or IV or recurrent endometrial cancer
* Poor curative potential with radiotherapy or surgery (alone or in combination)
* Measurable disease

  * At least one lesion accurately measured in at least one dimension

    * At least 20 mm by conventional techniques, including palpation, x-ray, CT scan, or MRI OR
    * At least 10 mm by spiral CT scan
  * Disease in a previously irradiated field as sole site of measurable disease allowed only if clear progression after completion of radiotherapy
* Estrogen receptor(ER)/progesterone receptor (PR) status of primary tumor required

  * ER/PR status of measurable tumor optional

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Granulocyte count at least 1,500/mm^3

Hepatic:

* Bilirubin normal
* SGPT no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 1.6 mg/dL

Cardiovascular:

* LVEF at least 50%
* No third-degree or complete heart block, unless pacemaker is in place
* Other conduction abnormalities or cardiac dysfunction allowed at the investigator's discretion
* No history of deep venous thrombosis
* No uncontrolled angina

Pulmonary:

* No history of pulmonary embolus

Other:

* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No concurrent medical illness that would preclude study
* No serious uncontrolled infection
* No serious peripheral neuropathy
* No circumstances that would preclude study compliance
* No sensitivity to E. coli-derived drug preparations

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy allowed

Chemotherapy:

* No prior cytotoxic chemotherapy, including chemotherapy for radiosensitization

Endocrine therapy:

* No prior hormonal therapy for endometrial cancer

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy involving the whole pelvis or more than 50% of the spine

Surgery:

* See Disease Characteristics

Other:

* Concurrent cardiac conduction-altering medications such as digitalis, beta blockers, or calcium channel blockers allowed at the investigator's discretion

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D. Bloss, MD, Study Chair — Washington University Siteman Cancer Center
Locations (50):
- United States (49):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - M.D. Anderson CCOP Research Base, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada